CLINICAL TRIAL: NCT02190513
Title: Prevalence of Eosinophilic Esophagitis in Children With Celiac Disease and Prevalence of Celiac Disease in Children With Eosinophilic Esophagitis in a Tertiary Community Hospital
Brief Title: Prevalence of Eosinophilic Esophagitis in Children With Celiac Disease
Status: Completed | Type: Observational
Sponsor: St. John Health System, Michigan (Other)
Responsible Party: Principal Investigator, Hernando Lyons, MD, tSection Chief of Pediatric Gastroenterology at St. John Hospital and Medical Center, St. John Health System, Michigan
Other Study IDs: SJ 0211-07
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Celiac Disease; Eosinophilic Esophagitis
MeSH Terms: conditions — Celiac Disease; Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Celiac disease (CD) and eosinophilic esophagitis (EE) are distinct diseases of the gastrointestinal tract with specific clinico-pathological characteristics. In recent years, in the literature, several children who underwent upper gastrointestinal endoscopy for suspected CD, which was confirmed histologically, were also found to have coexistent EE. There are reports of coexistent CD and EE. We would like to see the prevalence of EE in children with CD and the prevalence of CD in children with EE in our population, and to do so would like to review medical records. Our objectives are to determine if children with celiac disease have a high prevalence of eosinophilic esophagitis.and to determine if children with eosinophilic esophagitis have increased risk of developing celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Seen in the Pediatric Gastroenterology clinic at St. John Hospital & Medical Center during study time frame
* Age 2-21 years old
* Diagnosed with CD or EE or both based on the endoscopic and histopathological findings .

Exclusion Criteria:

* Gastroesophageal reflux diagnosed by PH probe.
* History of chemical ingestion

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children seen in the Pediatric Gastroenterology clinic at St. John Hospital & Medical Center and diagnosed with celiac disease or eosinophilic esophagitis or both based on the endoscopic and histopathological findings.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Review of histopathology reports of esophageal biopsies to record the number of eosinophils per high power field. | Retrospective chart review study, no contact made with patients, so no patient time is required, expected average of 2 years